CLINICAL TRIAL: NCT02804165
Title: Gene-virus Interactions Implicated in Type 1 Diabetes
Acronym: GENEVIR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-836
Record Dates: First submitted 2016-06-09; First posted 2016-06-17 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2017-05

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Enterovirus; Genetics; Gene-Virus interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Enterovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Target high-risk subjects or subpopulations for T1D (Other): Confirmation of the role of enteroviral infection in T1D and characterization of gene-enterovirus interactions should open up new avenues for understanding the pathogenesis of T1D and give clues on possible new therapeutic perspectives. Clinical applications might be further developed in order to extend the lag period might between positive autoantibodies detection and T1D age at onset in genetically predisposed subjects. This innovative project opens the door of the development of preventive therapy for T1D, as enterovirus vaccination.
  Interventions: Genetic: Enterovirus vaccination

INTERVENTIONS:
Genetic: Enterovirus vaccination — Enterovirus vaccination in genetically predisposed subjects having a high risk to develop type 1 diabetes.

SUMMARY:
Type 1 diabetes (T1D) is the most common endocrine disorder in children. In France, T1D prevalence is estimated to 12.2 per 100 000. Worldwide T1D incidence increased rapidly in the last decades, around 3% per year. T1D is caused by autoimmune destruction of pancreatic beta cells, leading to hyperglycaemia. T1D was recently associated an important loss in life expectancy compared with the general population. To date, the precise aetiology of T1D onset and the mechanisms involved in T1D remain unknown and no preventive treatment of T1D exists.

It is now well admitted that T1D results from a combined effect of genes, environmental factors and gene-environment interactions. Several genetic factors have been reported as associated to T1D, the most important being the human leukocyte antigen class II genes. Whole genome association studies suggested more than 50 T1D other susceptibility locus, but conferring individually a modest risk to develop T1D. Longitudinal studies demonstrated that only a low fraction of genetically predisposed subjects develop T1D and all these genetic factors cannot explain the increase in prevalence of T1D in the latter half of the 20th century, suggesting the implication of environmental factors.

Literature has accumulated a lot of evidence for the role of enterovirus in T1D. Several retrospective, prospective, post-mortem human studies, as well as animal studies, strongly suggest contribution of human enteroviruses to the pathogenesis of T1D. Enterovirus probably play a dual role in T1D, some enterovirus being associated with an increased risk of T1D and others with a protective effect. Interestingly, several T1D susceptibility loci are implicated in antiviral response. Epidemiologic and genetic approaches have led to new insights into T1D causation, but a collective explanation is still lacking.

The project aims at (1) demonstrating the gene-enterovirus interaction effect on T1D onset and (2) characterizing the "precipitating" effect of enterovirus on T1D by a follow-up study of T1D high-risk subjects (first degree unaffected relatives with positive autoantibodies to islet antigens).

A structural originality of this project is to perform a family-based study of gene-enterovirus interaction in T1D using innovative and robust methods. This project will be conducted in close collaboration between our INSERM unit, the Inter-regional network of paediatric diabetology, labelled biobanks (CBC Biotec of Hospices Civils de Lyon and CRB-LRB of Lariboisière' hospital at Paris), the Centre National de Référence des Enterovirus at Lyon and the Centre National de Génotypage at Evry.

The investigators will first conduct a 3-years pilot study (2016-2019), based on a sample of 250 nuclear families ascertained through a paediatric T1D proband in four centres. Families will be ascertained during the hospitalization of the proband at the time of T1D diagnosis. The study will be then extended to whole Inter-regional network of paediatric diabetology.

This research is a unique opportunity to explore further the implication of enterovirus and their interactions with genetic factors involved in T1D susceptibility and aims to target high-risk T1D subjects. This innovative project opens the door of the development of preventive therapy for T1D.

ELIGIBILITY:
Inclusion Criteria:

For Families :

For probands

* new-onset T1D (less than six months)
* aged between 2 and 15 years
* positive for T1D autoantibodies
* having at least one sib who accepts to participate to the study
* sign an informed consent form.

For relatives

* aged between 1 and 60 years
* having at least one sib (or child for parents) included in the study
* sign an informed consent form.

For unaffected T1D first degree relatives carrying antibodies to islet antigens:

* aged between 1 and 60 years
* being carrier of antibodies to islet antigens.
* having at least one sib (or child for parents) included in the study

Exclusion Criteria:

For Families :

* Adopted child
* For probands, being negative for T1D autoantibodies
* For probands, illness duration more than 6 months

For unaffected T1D first degree relatives carrying antibodies to islet antigens:

* being negative for T1D autoantibodies
* T1D patient

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Identification of gene-enterovirus interaction effect on T1D onset | 1 day
  The investigators choose to use a family-based approach in order to capture the underlying complexities of gene-environment interactions by identifying families with combinations of risk factors (genetic and enterovirus) that lead to disease expression. The gene-environment studies will be conducted for different candidate genes significantly associated with T1D. Families will be ascertained during the hospitalization of probands at the moment of T1D diagnosis. DNA, plasma, serum and stool samples will be collected for viral detection and genotyping. Gene-enterovirus effect will be estimated by using the "sibling-augmented case-only" approach based on logistic models.

SECONDARY OUTCOMES:
"Precipitating" effect of enterovirus infection on T1D. | 2 years
  Enterovirus infection "precipitating" effect will be tested by a survival analysis using the Cox semiparametric proportional hazards model, expressing the instantaneous hazard rate of T1D according to the status towards the enterovirus and covariates (age and gender).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Nicolino, MD, Principal Investigator — HCL
Locations (1):
- Hospices Civils de Lyon, Lyon, France